CLINICAL TRIAL: NCT06817707
Title: Evaluation of Urinary Dysfunction in CANVAS Patients
Acronym: UROCANVAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-AOIP-04
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cerebellar Ataxia; Neuropathy; Vestibular Areflexia
MeSH Terms: conditions — Cerebellar Ataxia; Bilateral Vestibulopathy | interventions — CANVAS syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Cerebellar Ataxia, Neuropathy, Vestibular Areflexia Syndrome (CANVAS) (Experimental)
  Interventions: Other: Evaluation of urinary dysfunction in patients with CANVAS

INTERVENTIONS:
Other: Evaluation of urinary dysfunction in patients with CANVAS — Urinary dysfunction will be evaluated with neurologic exam, interrogation, urinary dairy report, self-questionnaires, biologic analysis, Sudoscan and urological exams

SUMMARY:
The investigator wishes to evaluate the prevalence of urinary symptoms in patients diagnosed with Cerebellar Ataxia, Neuropathy, Vestibular Areflexia Syndrome (CANVAS).

As much as one third of patients living with CANVAS experience symptoms of urinary system dysfunction. The primary objective of this study is to evaluate the incidence of urinary symptoms in these patients, as well as the potential complications that might occur at the level of the upper and lower urinary system. The investigator also wishes to analyse the connection between the severity of the neurological deficits, the presence of dysautonomia and the presence of urinary dysfunction. To that end, the data collected in the study will concern : a detailed neurological examination including SARA (Scale for the assessement and rating of ataxia) scale assessement, laboratory tests of the renal function, dysautonomia tests with Sudoscan and research of orthostatic hypotension, urinary function questionnaires, dysautonomia questionnaire, urodynamic tests and urinary system ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more
* genetic confirmation of CANVAS (presence of pathogenic penta nucleotide expansion in both alleles of the replication factor C subunit 1(RFC1) gene or pathological penta nucleotide expansion in the heterozygous state associated with a truncating mutation on the second allele of the RFC1 gene)
* Able to undergo renovesical ultrasound and urinary flow measurement;
* Having given informed consent in writing;
* Negative pregnancy test for people on childbearing age;
* Social security affiliated

Exclusion Criteria:

* Presenting another urological pathology of base, not related to CANVAS;
* Having undergone a urological intervention within the 6 months preceding the screening visit;
* Presenting a condition that is incompatible with the proper conduct of the study as determined by the physician;
* Protected by law under guardianship or curators, or not able to participate in a clinical study pursuant to article L. 1121-16 of the French Public Health Code
* Pregnant or breastfeeding women for women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the prevalence of urinary dysfunctions in patients with CANVAS genetically confirmed | at inclusion
  The percentage of participants with urinary symptoms will be calculated by multiplying the number of participants with a USP (Urinary Symptom Profile) score greater than of equal to 1 by the total number of subjects included in the study, multiplied by 100. USP self-questionnaire was developped by the French Association of Urology. It aims to assess the symptoms of low urinary tract symptoms (LUTS) in men and women. It contains 13 items that assess stress urinary incontinence, bladder hyperreactivity and dysuria.

SECONDARY OUTCOMES:
Characterise the type of urinary dysfunctions | at inclusion
  To characterize the type of urinary dysfunctions (urinary incontinence, dysuria, bladder hyperactivity (urgent or pollakiuria)), we will use the answers to the USP (Urinary Symptom Profile) self-questionnaire. USP self-questionnaire was developped by the French Association of Urology. It aims to assess the symptoms of low urinary tract symptoms (LUTS) in men and women. It contains 13 items that assess stress urinary incontinence, bladder hyperreactivity and dysuria.
Characterise the severity of each type of urinary dysfunctions | at inclusion
  To characterize the degree of severity of urinary dysfunctions (mild, moderate, severe), we will use the answers to the IPSS (International Prostate Symptom Score) self-questionnaire. This questionnaire is a screening tool, which helps with the diagnosis and monitoring of symptoms of benign prostatic hypertrophy (BPH). It consists of 7 questions on urinary difficulties and one question on quality of life. Questions include: incomplete bladder emptying, frequency of urination, intermittent urination (stop and restart), urge to urinate (feeling "urgent"), low jet, effort to urinate (force or push), nycturia.
  Each question refers to the last month and has a score of 1 to 5, for a total of 35 points maximum.
  Patients can be classified according to the severity of symptoms: from 0 to 7 = low symptomatic; 8 to 19 = moderately symptomatic; from 20 to 35 = severe symptoms.
Characterise the impact of urinary dysfunctions on patient's quality of life | at inclusion
  To characterize the impact of urinary dysfunctions on patient's quality of life, we will use the SF-Qualiveen urological self-questionnaire. This questionnaire was developed to specifically and rapidly assess the impact on quality of life of urinary disorders in patients with a neurological bladder. Its initial validation was performed in patients with multiple sclerosis. This rapid form of the Qualiveen scale has 8 items evaluating 4 domains: discomfort, constraints, fears and patient experience. Each item is rated from 0 to 4
Assess the prevalence of different types of urinary dysfunctions | at inclusion
  To calculate the prevalence of each type of urinary dysfunctions (urinary incontinence, dysuria, bladder hyperactivity (urgent or pollakiuria)), the percentage of participants with each type of impairment will be calculated as the ratio between the number of subjects in each group of impairment and the total number of participants with a USP score greater than or equal to 1, multiplied by 100.
Assess the prevalence of biological complications in the upper urinary tract | at inclusion
  To calculate the prevalence of biological complications in the upper urinary tract, the percentage of subjects with abnormal renal function at the biological balance will be calculated by the ratio of the number of subjects with glomerular filtration rate (GFR) < 90 mL/min/1,73 m2 and the total number of participants with a USP score greater than or equal to 1, multiplied by 100.
Assess the prevalence of structural complications in the upper urinary tract | within 6 months after inclusion
  To calculate the prevalence of structural complications in the upper urinary tract, the percentage of subjects with structural abnormalities of the urinary system will be calculated by the ratio of the number of subjects with pyelocalicial dilation, renal lithiasis or abnormal bladder wall on renal ultrasound and the total number of participants with a USP score greater than or equal to 1, multiplied by 100.
Assess prevalence of urinary flow malfunction | within 6 months after inclusion
  To calculate the prevalence of urinary flow malfunction, the percentage of subjects with functional urinary anomalies will be calculated by the ratio of the number of subjects with a deviation from the bladder emptying curve, or a maximum flow rate < 15 mL at urinary flow, or a post-micturition residue greater than 100 mL and the total number of participants with USP greater than or equal to 1, multiplied by 100.
Assess prevalence of dysautonomia | at inclusion
  To assess the prevalence of dysautonomia, the percentage of subjects with dysautonomia will be calculated by the ratio of participants with a positive Sudoscan or orthostatic hypotension test and the total number of participants, multiplied by 100.
Assess the prevalence of dysautonomia symptoms | at inclusion
  To calculate the prevalence of dysautonomia symptoms, the percentage of subjects with dysautonomia symptoms will be calculated as the ratio between the number of subjects with an abnormal response to the SCOPA-AUT (Scales for outcome in Parkinson's disease - Autonomic dysfunction) questionnaire and the total number of participants, multiplied by 100. The SCOPA-AUT is a validated scale developed to assess symptoms of dysautonomia in patients with Parkinson's disease and multisystemic atrophy. It allows to evaluate the symptoms of digestive, urinary, sexual, thermoregulatory, pupillary and cardiovascular dysfunction. It is composed of 26 questions. Each question refers to the last month and has a score of 1 to 4 or 5.
Assess the relationship between urinary dysfunction and presence of dysautonomia | at inclusion
  To assess the association between urinary dysfunction and dysautonomia, we will compare the percentage of participants with a UPS score greater than or equal to 1 among participants who have dysautonomia (following the SCOPA-AUT questionnaire, the SUDOSCAN test or the search for orthostatic hypotension), and the percentage of participants with a USP score greater than or equal to 1 among participants without dysautonomia.
Assess the relationship between severity of neurological dysfunction and dysautonomia | at inclusion
  To assess the relationship between severity of neurological dysfunction and dysautonomia, we will calculate the SARA (Scale for the assessement and rating of ataxia) score for each participant and divide patients into 3 subgroups: Group 1 (SARA score < 15), Group 2 (SARA score between 15 - 25) and Group 3 (SARA score > 25). The SARA score was developed to evaluate the various deficits resulting from cerebellum dysfunction. It is divided into 8 categories with a cumulative score of 0 (without ataxia) to 40 (the most severe form of ataxia): walking, standing, sitting, speaking, finger hunting, nose test - quick alternate hand movements, heel slip - ankle. For items 5 to 8, the assessment is done bilaterally and then the average value is calculated to obtain the final score.
  We will then calculate and compare the percentage of subjects with dysautonomia (following SCOPA AUT questionnaire, SUDOSCAN test or search for orthostatic hypotension) in each SARA score group.
Assess the relationship between urinary dysfunction and severity of neurological dysfunction | at inclusion
  To assess the relationship between urinary dysfunction and severity of neurological dysfunction, we will calculate and compare the percentage of subjects with urological symptoms or a USP score greater than or equal to 1 in each SARA score group.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nice University Hospital, Nice, Alpes Maritimes
  - Montpellier University hospital, Montpellier, Hérault
  - Lille University Hospital, Lille, Nord

IPD SHARING:
Plan to Share IPD: No